CLINICAL TRIAL: NCT02485938
Title: A Randomized, Open-label Study of the Safety and Efficacy of Multi- Vessel Intracoronary Delivery of Allogeneic Cardiosphere-Derived Cells in Patients With Cardiomyopathy Secondary to Duchenne Muscular Dystrophy
Brief Title: HOPE-Duchenne (Halt cardiomyOPathy progrEssion in Duchenne)
Acronym: HOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capricor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAP-1002-DMD-01
Record Dates: First submitted 2015-06-19; First posted 2015-06-30 (Estimated); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Duchenne Muscular Dystrophy; Cardiomyopathy
Keywords: Duchenne Muscular Dystrophy; Cardiomyopathy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Allogeneic Cardiosphere-Derived Cells (CAP-1002) (Experimental): CAP-1002 is an investigational product consisting of allogeneic cardiosphere-derived cells (CDCs). All subjects assigned to the active treatment arm will receive an intended total dose of 75 million (M) CAP-1002 cells infused as 25M cells into each of the three left ventricle cardiac territories (anterior, lateral, inferior/posterior). If any of the three coronary arteries are deemed by the infusing Investigator to supply less than 30% of the left ventricular myocardium, the infusing Investigator may choose to infuse only 12.5M cells into that coronary artery or arteries. Therefore the full dose of CAP-1002 delivered may range from 50M cells to 75M cells provided that all three arteries are infused.
  Interventions: Drug: Allogeneic Cardiosphere-Derived Cells (CAP-1002)
- Usual Care (No Intervention): Subjects randomized to receive usual care will continue to be cared for and treated in whatever manner the investigator deems most appropriate for the subject on an ongoing basis, and will receive no infusion.

INTERVENTIONS:
Drug: Allogeneic Cardiosphere-Derived Cells (CAP-1002) — Intracoronary delivery of Allogeneic Cardiosphere-Derived Cells (CAP-1002)
  Other Names: CAP-1002
  Arms: Allogeneic Cardiosphere-Derived Cells (CAP-1002)

SUMMARY:
Male participants with cardiomyopathy secondary to Duchenne muscular dystrophy (DMD) meeting all inclusion and no exclusion criteria will be randomized. All participants will be at least 12 years of age. They will be randomized in a 1:1 manner to either intracoronary infusion of CAP-1002 in three coronary arteries supplying the three major cardiac territories of the left ventricle of the heart (anterior, lateral, inferior/posterior) or usual care. In the active treatment arm, all three major cardiac territories will be treated (infused) during a single procedure in an open-label fashion.

DETAILED DESCRIPTION:
Approximately 24, and not more than 30, participants will be randomized into the study, in two sequential enrollment groups. Safety data from Group 1 will undergo a Data Safety Monitoring Board (DSMB) review prior to initiation of enrollment for Group 2.

The first 6-8 randomized participants will comprise Group 1, and will include a minimum of 3 participants completing intracoronary infusion with CAP-1002. The DSMB will conduct a review of interim safety data through 72 hours post-Day 0 for at least 3 infused participants and for at least 6 participants overall.

Enrollment of Group 2 will begin per DSMB recommendations following their review of the 72 hour safety data from Group 1. Group 2 will include approximately 18 participants. Screening and randomization will continue until at total of 12 participants are infused with CAP 1002 or 30 participants are randomized into the study, whichever comes first.

All participants assigned to the active treatment arm will receive an intended total dose of up to 75 million (M) CAP-1002 cells infused as 25M cells into each of the three left ventricle cardiac territories (anterior, lateral, inferior/posterior).

Participants randomized to receive usual care will continue to be cared for and treated in whatever manner the investigator deems most appropriate for the participant on an ongoing basis, and will receive no infusion.

Randomization will take place within 30 days of the first screening procedure. After completion of the screening procedures, eligible participants randomized to active treatment arm will receive CAP-1002 administered via intracoronary infusion on Day 0. Day 0 for eligible participants randomized to the usual care arm will occur 7 days after the date of randomization. All randomized participants will have a follow-up telephone call on Study Day 3, and study visits at Weeks 2 and 6, and at Months 3, 6 and 12 post Day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants 18 years of age or older must be able to provide informed consent and follow up with protocol procedures. Male participants at least 12 years of age but younger than 18 years of age must be able to provide assent with parent or guardian providing permission for study participation. Only male participants will be randomized into this study.
2. Documented diagnosis of Duchenne Muscular Dystrophy by genetic mutation analysis.
3. Cardiomyopathy with left ventricular scar by late gadolinium enhancement (LGE) in at least 4 segments as assessed by contrast-enhanced MRI and EF >35% at the time of screening.
4. Use of evidence based medical-therapy in accordance with the "DMD Care Considerations Working Group" guidelines for the management of DMD, for at least three months prior to signing the consent form (or, providing assent) or documented contraindication or intolerance or patient preference.
5. Participants must be taking systemic glucocorticoids for at least six months prior to screening.
6. Participants must be 12 years of age or older at time of screening
7. Participants must be appropriate candidates for cardiac catheterization and intracoronary infusion of CAP-1002, in the judgement of the site's interventional cardiologist.

Exclusion Criteria:

1. Therapy with intravenous inotropic or vasoactive medications at the time of screening.
2. Inability to undergo cardiac catheterization and/or MRI without general anesthesia.
3. Immunologic incompatibility with all available Master Cell Banks (MCBs) by single-antigen bead (SAB) serum antibody profiling.
4. Planned or likely major surgery in the next 12 months after planned randomization.
5. Left Ventricular Assist Devices (LVAD) or those subjects actively in the process of acquiring a LVAD.
6. Contraindication to cardiac MRI.
7. Known hypersensitivity to contrast agents.
8. Estimated glomerular filtration rate (GFR) <60 mL/min, as calculated by the CKD-EPI cystatin C equation (Inker, Schmid et al. 2012).
9. Active infection not responsive to treatment.
10. Active systemic allergic reaction(s), connective tissue disease or autoimmune disorder(s).
11. History of cardiac tumor or cardiac tumor demonstrated on screening MRI.
12. History of previous stem cell therapy.
13. History of use of medications listed in Appendix 3 within 3 months prior to signing the Inform Consent Form / Assent through completion of the study infusion.
14. Known moderate-to-severe aortic stenosis/insufficiency or severe mitral stenosis/regurgitation.
15. Current active alcohol or drug abuse.
16. Known history of Human Immunodeficiency Virus (HIV) infection.
17. Known history of chronic viral hepatitis.
18. Abnormal liver function (alanine aminotransferase (ALT)/aspartate aminotransferase (AST) >10 times the upper reference range) and/or abnormal hematology (hematocrit <25%, White Blood Cells <3000 μl, platelets <100,000 μl) studies without a reversible, identifiable cause.
19. Known hypersensitivity to bovine products.
20. Known hypersensitivity to dimethyl sulfoxide (DMSO).
21. Uncontrolled diabetes (HbA1c >9.0).
22. Inability to comply with protocol-related procedures, including required study visits.
23. Any condition or other reason that, in the opinion of the Investigator or Medical Monitor, would render the subject unsuitable for the study.
24. Currently receiving investigational treatment on another clinical study or expanded access protocol, including any of the following:

    * Received investigational intervention within 30 days prior to randomization
    * Treatment and/or an incomplete follow-up to treatment with any investigational cell based therapy within 6 months prior to randomization
    * Active participation in other research therapy for cardiovascular repair/regeneration

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Awadalla, Study Director — Capricor Inc.
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants at 3 active sites between 07 January 2016 to 14 September 2017.
Pre-assignment Details: Participants were randomized in 1:1 ratio to receive either Allogeneic Cardiosphere-Derived Cells (CAP-1002) or usual care. Usual care participants were considered as a reference comparator group and received no treatment.
Groups:
- Usual Care: Participants randomized to receive usual care continued to be cared for and treated in the manner the investigator deemed most appropriate for the participant on an ongoing basis and received no infusion.
- CAP-1002: Participants received an intended total dose of 75 million (M) cardiosphere-derived cells (CDCs) infused as 25M cells into each of the three main coronary arteries supplying the anterior, lateral and inferior/posterior cardiac territories during a single, intracoronary procedure on Day 0 and were followed up for 12 months post-infusion.
Period: Overall Study
Arm/Group | Usual Care | CAP-1002
Started | 12 | 13
Completed | 10 | 13
Not Completed | 2 | 0
Not completed — Withdrawal of consent | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population that included all participants who received CAP-1002 treatment on Day 0 and all participants in the usual care treatment group who remained in study as of the reference time point.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | CAP-1002 | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.9 (2.75) | 18.7 (3.50) | 17.8 (3.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 11 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Any of the Adjudicated Events
Description: Adjudicated Events reported included: New thrombolysis in myocardial infarction (TIMI) flow 0-2 or TIMI myocardial perfusion grade (TMPG) 0-2noted immediately following infusion and persisting greater than (>) 3 minutes, despite intracoronary vasodilator administration; sudden unexpected death within 72 hours of intracoronary infusion; and Major adverse cardiac event (MACE) within 72 hours of intracoronary infusion, including death, non-fatal myocardial infarction and hospitalization for cardiovascular event (including heart failure hospitalizations).
Time Frame: Within 72 hours post-infusion
Population: Analysis was performed on safety population that included all participants who received CAP-1002 treatment on Day 0 and all participants in the usual care treatment group who remained in study as of the reference time point. Participants were summarized and analyzed per treatment actually received, regardless of their randomization assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
Participants
  TIMI 0-2 | 0 | 0
  Sudden unexpected death | 0 | 0
  MACE | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily had to have causal relationship with treatment. TEAEs were defined as AEs that occurred or worsened in severity between the first dose of the investigational medicinal product (IMP) until the end of study. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalisation or prolongation of existing hospitalisation, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: Up to Month 12 post-infusion
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
Participants
  TEAEs | 10 | 12
  SAEs | 1 | 3

3. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters (Chloride, Potassium and Sodium) at Month 6 and Month 12
Description: Clinical chemistry parameters assessed were chloride, potassium and sodium.
Time Frame: Baseline, Month 6 and Month 12
Population: Analysis was performed on safety population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
millimoles per liter (mmol/L)
  Chloride: Baseline | 100.9 (2.54) | 102.7 (3.52)
  Chloride: Change at Month 6: number analyzed (Participants) | 11 | 12
  Chloride: Change at Month 6 | -0.4 (2.46) | -0.8 (4.09)
  Chloride: Change at Month 12: number analyzed (Participants) | 10 | 13
  Chloride: Change at Month 12 | 0.2 (2.53) | -0.9 (3.95)
  Potassium: Baseline | 4.28 (0.252) | 4.00 (0.356)
  Potassium: Change at Month 6: number analyzed (Participants) | 11 | 13
  Potassium: Change at Month 6 | -0.15 (0.342) | 0.22 (0.286)
  Potassium: Change at Month 12: number analyzed (Participants) | 10 | 13
  Potassium: Change at Month 12 | -0.08 (0.531) | 0.31 (0.362)
  Sodium: Baseline | 138.7 (2.23) | 140.2 (2.51)
  Sodium: Change at Month 6: number analyzed (Participants) | 11 | 13
  Sodium: Change at Month 6 | -0.3 (2.90) | -1.5 (3.15)
  Sodium: Change at Month 12: number analyzed (Participants) | 10 | 13
  Sodium: Change at Month 12 | 0.3 (1.83) | -1.2 (2.83)

4. Primary Outcome: Change From Baseline in Clinical Laboratory Parameter - Albumin at Month 6 and Month 12
Description: Clinical chemistry parameter assessed was albumin.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
grams per deciliter
  Baseline | 4.48 (0.266) | 3.87 (0.417)
  Change at Month 6: number analyzed (Participants) | 11 | 13
  Change at Month 6 | -0.09 (0.181) | 0.36 (0.500)
  Change at Month 12: number analyzed (Participants) | 10 | 13
  Change at Month 12 | -0.02 (0.199) | 0.32 (0.402)

5. Primary Outcome: Change From Baseline in Clinical Laboratory Parameter - Glucose at Month 6 and Month 12
Description: Clinical chemistry parameter assessed was glucose.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
milligrams per deciliter
  Baseline | 87.1 (8.20) | 89.5 (9.58)
  Change at Month 6: number analyzed (Participants) | 11 | 13
  Change at Month 6 | 2.1 (13.78) | 12.3 (20.56)
  Change at Month 12: number analyzed (Participants) | 10 | 13
  Change at Month 12 | -4.1 (12.44) | 6.8 (15.00)

6. Primary Outcome: Change From Baseline in Hematological Parameters (Platelets, White Blood Cells, Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils) at Month 6 and Month 12
Description: Hematological parameters assessed were: platelets, white blood cells, basophils, eosinophils, lymphocytes, monocytes and neutrophils.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
10^3 cells per microliter
  Platelets: Baseline | 357.9 (68.36) | 318.6 (53.63)
  Platelets: Change at Month 6: number analyzed (Participants) | 11 | 12
  Platelets: Change at Month 6 | -24.5 (51.25) | 40.4 (45.39)
  Platelets: Change at Month 12: number analyzed (Participants) | 9 | 13
  Platelets: Change at Month 12 | -26.0 (45.72) | 24.0 (43.10)
  White Blood Cells: Baseline | 9.83 (3.001) | 10.57 (3.947)
  White Blood Cells: Change at Month 6: number analyzed (Participants) | 11 | 12
  White Blood Cells: Change at Month 6 | 1.11 (4.010) | 0.81 (2.606)
  White Blood Cells: Change at Month 12: number analyzed (Participants) | 9 | 12
  White Blood Cells: Change at Month 12 | 0.42 (2.348) | -0.28 (1.556)
  Basophils: Baseline | 0.033 (0.0218) | 0.060 (0.1052)
  Basophils: Change at Month 6: number analyzed (Participants) | 11 | 12
  Basophils: Change at Month 6 | -0.004 (0.0196) | -0.033 (0.1064)
  Basophils: Change at Month 12: number analyzed (Participants) | 9 | 12
  Basophils: Change at Month 12 | 0.012 (0.0264) | -0.040 (0.1197)
  Eosinophils: Baseline | 0.136 (0.1154) | 0.171 (0.1848)
  Eosinophils: Change at Month 6: number analyzed (Participants) | 11 | 12
  Eosinophils: Change at Month 6 | -0.005 (0.1296) | -0.073 (0.1515)
  Eosinophils: Change at Month 12: number analyzed (Participants) | 9 | 12
  Eosinophils: Change at Month 12 | 0.067 (0.1742) | -0.078 (0.1366)
  Lymphocytes: Baseline | 2.793 (1.0429) | 3.381 (1.5423)
  Lymphocytes: Change at Month 6: number analyzed (Participants) | 11 | 12
  Lymphocytes: Change at Month 6 | -0.595 (1.1509) | -0.918 (1.9381)
  Lymphocytes: Change at Month 12: number analyzed (Participants) | 9 | 12
  Lymphocytes: Change at Month 12 | 0.771 (1.5711) | -0.393 (1.5501)
  Monocytes: Baseline | 0.413 (0.1707) | 0.705 (0.2608)
  Monocytes: Change at Month 6: number analyzed (Participants) | 11 | 12
  Monocytes: Change at Month 6 | -0.082 (0.2248) | -0.273 (0.4337)
  Monocytes: Change at Month 12: number analyzed (Participants) | 9 | 12
  Monocytes: Change at Month 12 | 0.009 (0.2036) | -0.284 (0.3238)
  Neutrophils: Baseline | 6.475 (2.7169) | 6.198 (2.9121)
  Neutrophils: Change at Month 6: number analyzed (Participants) | 11 | 12
  Neutrophils: Change at Month 6 | 1.783 (4.2366) | 2.153 (3.4484)
  Neutrophils: Change at Month 12: number analyzed (Participants) | 9 | 12
  Neutrophils: Change at Month 12 | -0.451 (2.5038) | 0.566 (1.9689)

7. Primary Outcome: Change From Baseline in Hematological Parameter - Hemoglobin at Month 6 and Month 12
Description: Hematological parameter assessed was hemoglobin.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
grams per deciliter
  Baseline | 14.48 (0.651) | 13.76 (1.254)
  Change at Month 6: number analyzed (Participants) | 11 | 12
  Change at Month 6 | -0.05 (1.054) | 0.05 (0.458)
  Change at Month 12: number analyzed (Participants) | 9 | 13
  Change at Month 12 | -0.13 (1.288) | 0.29 (0.808)

8. Primary Outcome: Change From Baseline in Hematological Parameter - Red Blood Cells at Month 6 and Month 12
Description: Hematological parameter assessed was red blood cells.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
10^6 cells per microliter
  Baseline | 5.01 (0.309) | 4.68 (0.414)
  Change at Month 6: number analyzed (Participants) | 11 | 12
  Change at Month 6 | -0.05 (0.372) | 0.20 (0.286)
  Change at Month 12: number analyzed (Participants) | 9 | 13
  Change at Month 12 | -0.07 (0.415) | 0.23 (0.340)

9. Primary Outcome: Change From Baseline in Vital Signs - Blood Pressure at Month 6 and Month 12
Description: Vital signs assessed were systolic and diastolic blood pressure.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
millimeters of mercury
  Systolic Blood Pressure: Baseline | 111.3 (12.29) | 113.7 (12.72)
  Systolic Blood Pressure: Change at Month 6: number analyzed (Participants) | 11 | 13
  Systolic Blood Pressure: Change at Month 6 | 2.3 (18.70) | -2.1 (11.98)
  Systolic Blood Pressure: Change at Month 12: number analyzed (Participants) | 10 | 13
  Systolic Blood Pressure: Change at Month 12 | -0.3 (9.66) | 2.8 (17.67)
  Diastolic Blood Pressure: Baseline | 65.9 (11.92) | 66.7 (14.12)
  Diastolic Blood Pressure: Change at Month 6: number analyzed (Participants) | 11 | 13
  Diastolic Blood Pressure: Change at Month 6 | -0.3 (10.49) | 0.1 (14.52)
  Diastolic Blood Pressure: Change at Month 12: number analyzed (Participants) | 10 | 13
  Diastolic Blood Pressure: Change at Month 12 | 3.5 (8.92) | 1.5 (14.79)

10. Primary Outcome: Change From Baseline in Vital Signs - Heart Rate at Month 6 and Month 12
Description: Vital signs assessed was heart rate.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
beats per minute
  Baseline | 90.8 (9.18) | 87.1 (14.71)
  Change at Month 6: number analyzed (Participants) | 11 | 13
  Change at Month 6 | -3.0 (13.42) | 4.8 (12.43)
  Change at Month 12: number analyzed (Participants) | 10 | 13
  Change at Month 12 | -0.2 (13.39) | 4.4 (11.24)

11. Primary Outcome: Change From Baseline in Vital Signs - Respiratory Rate at Month 6 and Month 12
Description: Vital signs assessed was respiratory rate.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
breaths per minute
  Baseline | 17.3 (2.27) | 16.3 (2.81)
  Change at Month 6: number analyzed (Participants) | 11 | 13
  Change at Month 6 | -0.5 (1.75) | 0.3 (3.71)
  Change at Month 12: number analyzed (Participants) | 10 | 13
  Change at Month 12 | 0.0 (2.00) | 0.8 (4.21)

12. Primary Outcome: Change From Baseline in Vital Signs - Temperature at Month 6 and Month 12
Description: Vital signs assessed was temperature.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: celsius
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
celsius
  Baseline: number analyzed (Participants) | 11 | 13
  Baseline | 36.79 (0.362) | 36.68 (0.360)
  Change at Month 6: number analyzed (Participants) | 10 | 13
  Change at Month 6 | -0.13 (0.490) | 0.18 (0.545)
  Change at Month 12: number analyzed (Participants) | 9 | 13
  Change at Month 12 | -0.09 (0.276) | 0.05 (0.609)

13. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Cardiac Physical Examinations at Month 6 and Month 12
Description: Cardiac physical examination parameters assessed were: jugular vein distension, edema, heart sounds, murmur, breath sounds.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
Participants
  Jugular Vein Distension: Month 6: number analyzed (Participants) | 11 | 13
  Jugular Vein Distension: Month 6 | 0 | 0
  Jugular Vein Distension: Month 12: number analyzed (Participants) | 10 | 13
  Jugular Vein Distension: Month 12 | 0 | 0
  Edema: Month 6: number analyzed (Participants) | 11 | 13
  Edema: Month 6 | 1 | 1
  Edema: Month 12: number analyzed (Participants) | 10 | 13
  Edema: Month 12 | 0 | 1
  Heart Sounds: Month 6: number analyzed (Participants) | 11 | 13
  Heart Sounds: Month 6 | 1 | 0
  Heart Sounds: Month 12: number analyzed (Participants) | 10 | 13
  Heart Sounds: Month 12 | 1 | 1
  Murmur: Month 6: number analyzed (Participants) | 11 | 13
  Murmur: Month 6 | 0 | 0
  Murmur: Month 12: number analyzed (Participants) | 10 | 13
  Murmur: Month 12 | 0 | 0
  Breath Sounds: Month 6: number analyzed (Participants) | 11 | 13
  Breath Sounds: Month 6 | 1 | 0
  Breath Sounds: Month 12: number analyzed (Participants) | 10 | 13
  Breath Sounds: Month 12 | 1 | 2

14. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters (QRS Duration, PR, QT, QTc and QT Interval) at Month 6 and Month 12
Description: ECG parameters assessed were: PR Interval, QRS Duration, QT Interval, QTc interval and QT interval.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
millisecond
  PR Interval: Baseline | 116.2 (41.23) | 129.2 (21.31)
  PR Interval: Change at Month 6: number analyzed (Participants) | 11 | 13
  PR Interval: Change at Month 6 | 8.7 (37.02) | -2.8 (7.67)
  PR Interval: Change at Month 12: number analyzed (Participants) | 10 | 13
  PR Interval: Change at Month 12 | 8.3 (44.40) | 1.0 (12.58)
  QRS Duration: Baseline | 92.7 (8.11) | 91.3 (10.03)
  QRS Duration: Change at Month 6: number analyzed (Participants) | 11 | 13
  QRS Duration: Change at Month 6 | -0.8 (7.25) | 4.5 (7.58)
  QRS Duration: Change at Month 12: number analyzed (Participants) | 10 | 13
  QRS Duration: Change at Month 12 | 4.1 (9.53) | 4.5 (6.04)
  QT Interval: Baseline | 350.6 (18.76) | 348.9 (21.55)
  QT Interval: Change at Month 6: number analyzed (Participants) | 11 | 13
  QT Interval: Change at Month 6 | 4.4 (16.07) | -3.2 (18.91)
  QT Interval: Change at Month 12: number analyzed (Participants) | 10 | 13
  QT Interval: Change at Month 12 | 11.7 (23.90) | -0.2 (18.21)
  QTc Interval: Baseline | 419.6 (25.25) | 423.7 (23.60)
  QTc Interval: Change at Month 6: number analyzed (Participants) | 11 | 13
  QTc Interval: Change at Month 6 | 6.5 (11.84) | -5.8 (23.45)
  QTc Interval: Change at Month 12: number analyzed (Participants) | 10 | 13
  QTc Interval: Change at Month 12 | 8.4 (6.42) | 1.2 (27.23)

15. Primary Outcome: Change From Baseline in Electrocardiogram Parameter - Ventricular Rate at Month 6 and Month 12
Description: ECG parameter assessed was ventricular rate; which depends on the degree of atrioventricular conduction.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 12 | 13
beats per minute
  Baseline | 87.8 (11.95) | 89.8 (14.43)
  Change at Month 6: number analyzed (Participants) | 11 | 13
  Change at Month 6 | 0.8 (7.11) | 1.2 (14.66)
  Change at Month 12: number analyzed (Participants) | 10 | 13
  Change at Month 12 | -1.8 (11.11) | 2.2 (14.62)

16. Other Pre Specified Outcome: Absolute Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Month 6 and 12
Description: LVEF is the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume). LVEF expressed as percentage ejection fraction was assessed by magnetic resonance imaging. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percentage ejection fraction
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percentage ejection fraction
  Month 6 | 0.74 (5.497) | 1.07 (3.376)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | 0.624 (4.396) | -0.35 (2.703)

17. Other Pre Specified Outcome: Percent Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Month 6 and 12
Description: LVEF is the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume). Percent change in LVEF was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent change
  Month 6 | 2.35 (10.456) | 2.44 (7.301)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | 1.88 (8.830) | -0.88 (5.580)

18. Other Pre Specified Outcome: Absolute Change From Baseline in Left Ventricular End Diastolic Volume (LVEDV) at Month 6 and 12
Description: LVEDV is the amount of blood in the heart's left ventricle just before the heart contracts. LVEDV was assessed by magnetic resonance imaging. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
milliliters (mL)
  Month 6 | 3.44 (14.311) | 0.14 (8.538)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | 3.21 (12.309) | 6.16 (11.655)

19. Other Pre Specified Outcome: Percent Change From Baseline in Left Ventricular End Diastolic Volume (LVEDV) at Month 6 and 12
Description: LVEDV is the amount of blood in the heart's left ventricle just before the heart contracts. Percent change in LVEDV was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent change
  Month 6 | 2.13 (9.851) | -0.28 (7.246)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | 1.86 (9.567) | 3.91 (8.479)

20. Other Pre Specified Outcome: Absolute Change From Baseline in Left Ventricular End Systolic Volume (LVESV) at Month 6 and 12
Description: LVESV is the amount of blood remaining in the ventricle at the end of systole, after the heart has contracted. LVESV was assessed by magnetic resonance imaging. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
mL
  Month 6 | 0.60 (8.800) | -0.79 (5.869)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | 1.29 (7.132) | 4.51 (8.000)

21. Other Pre Specified Outcome: Percent Change From Baseline in Left Ventricular End Systolic Volume (LVESV) at Month 6 and 12
Description: LVESV is the amount of blood remaining in the ventricle at the end of systole, after the heart has contracted. Percent change in LVESV was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent change
  Month 6 | 0.96 (10.987) | -2.12 (10.558)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | 1.17 (12.706) | 4.43 (9.881)

22. Other Pre Specified Outcome: Absolute Change From Baseline in LV Late Gadolinium Enhancement (LGE) Scar Tissue Mass at Month 6 and 12
Description: Late gadolinium enhancement is a technique used in cardiac MRI for cardiac tissue characterization, in particular, the assessment of myocardial scar formation and regional myocardial fibrosis. LV LGE scar tissue mass in grams was assessed by cardiac MRI. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
grams
  Month 6 | 1.07 (2.564) | 0.29 (3.038)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | 0.99 (5.163) | -0.15 (3.302)

23. Other Pre Specified Outcome: Percent Change From Baseline in LV Late Gadolinium Enhancement (LGE) Scar Tissue Mass at Month 6 and 12
Description: Late gadolinium enhancement is a technique used in cardiac MRI for cardiac tissue characterization, in particular, the assessment of myocardial scar formation and regional myocardial fibrosis. Percent change in LV LGE scar tissue mass was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent change
  Month 6 | 9.42 (14.056) | -0.39 (19.032)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | 10.86 (23.17) | -2.81 (19.557)

24. Other Pre Specified Outcome: Absolute Change From Baseline in Left Ventricular (LV) Late Gadolinium Enhancement (LGE) at Month 6 and 12
Description: Late gadolinium enhancement is a technique used in cardiac MRI for cardiac tissue characterization, in particular, the assessment of myocardial scar formation and regional myocardial fibrosis. Improvement in infarct size as a percent of LV mass was assessed by magnetic resonance imaging and reported in this outcome measure.
Time Frame: Baseline, Month 6 and 12
Population: Analysis was performed on modified intent-to-treat (mITT) population that included all participants who received CAP-1002 treatment on Day 0 and all participants in the usual care treatment group who remained in study as of the reference time point and had at least one post-baseline observation. Participants were summarized and analyzed per treatment actually received, regardless of their randomization assignment. 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percent of LV mass
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent of LV mass
  Month 6 | -0.53 (2.865) | -1.11 (1.630)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | -0.09 (5.472) | -1.35 (1.778)

25. Other Pre Specified Outcome: Percent Change From Baseline in LV Late Gadolinium Enhancement (LGE) at Month 6 and 12
Description: Late gadolinium enhancement is a technique used in cardiac MRI for cardiac tissue characterization, in particular, the assessment of myocardial scar formation and regional myocardial fibrosis. Percent improvement in infarct size defined by scar as a percent of LV mass was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent change
  Month 6 | -0.23 (11.482) | -5.09 (8.480)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | 4.76 (22.253) | -7.14 (10.298)

26. Other Pre Specified Outcome: Absolute Change From Baseline in Circumferential Strain at Month 6 and 12
Description: Circumferential strain represents the change in length (shortening in systole, represented as a negative strain value) of the myocardium along the circumferential axis of the LV as viewed in the short axis. Improvement in Circumferential Strain was expressed in percentage and was assessed by cardiac MRI.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percentage circumferential strain
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percentage circumferential strain
  Month 6 | -0.586 (2.9542) | -0.616 (1.7732)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | -0.173 (2.6342) | -0.707 (2.4454)

27. Other Pre Specified Outcome: Percent Change From Baseline in Circumferential Strain at Month 6 and 12
Description: Circumferential strain represents the change in length (shortening in systole, represented as a negative strain value) of the myocardium along the circumferential axis of the LV as viewed in the short axis; and was assessed by cardiac MRI. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent change
  Month 6 | -4.62 (24.100) | -6.40 (15.198)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | -1.50 (21.755) | -9.17 (24.823)

28. Other Pre Specified Outcome: Change From Baseline in Function of the Region Receiving CAP-1002 Therapy at Month 6 and 12
Description: The regions assessed of the heart were: Anterior, Lateral, Inferior and Septal. Tissue mass recovery in the function of region receiving therapy expressed as change from baseline was assessed by magnetic resonance imaging. Change was calculated as: post-baseline value - baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent
  Anterior: Month 6 | -8.20 (14.763) | 2.72 (14.256)
  Anterior: Month 12: number analyzed (Participants) | 10 | 13
  Anterior: Month 12 | 2.28 (10.342) | 5.17 (11.757)
  Lateral: Month 6 | -2.73 (11.487) | 5.21 (12.704)
  Lateral: Month 12: number analyzed (Participants) | 10 | 13
  Lateral: Month 12 | 3.94 (13.011) | 6.16 (8.353)
  Inferior: Month 6 | -4.52 (9.706) | 7.78 (11.470)
  Inferior: Month 12: number analyzed (Participants) | 10 | 13
  Inferior: Month 12 | -2.74 (9.739) | 7.98 (12.494)
  Septal: Month 6 | -0.59 (14.530) | 1.01 (13.728)
  Septal: Month 12: number analyzed (Participants) | 10 | 13
  Septal: Month 12 | 0.86 (12.177) | 4.94 (11.981)

29. Other Pre Specified Outcome: Percent Change From Baseline in Function of the Region Receiving CAP-1002 Therapy at Month 6 and 12
Description: The regions assessed of the heart were: Anterior, Lateral, Inferior and Septal. Tissue mass recovery in the function of region receiving therapy expressed as percent change from baseline was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value - Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent change
  Anterior: Month 6 | -14.12 (24.899) | 16.25 (46.546)
  Anterior: Month 12: number analyzed (Participants) | 10 | 13
  Anterior: Month 12 | 12.75 (32.836) | 21.76 (44.713)
  Lateral: Month 6 | -4.54 (35.009) | 24.50 (51.156)
  Lateral: Month 12: number analyzed (Participants) | 10 | 13
  Lateral: Month 12 | 25.49 (63.231) | 28.22 (40.267)
  Inferior: Month 6 | -8.78 (27.679) | 31.19 (46.995)
  Inferior: Month 12: number analyzed (Participants) | 10 | 13
  Inferior: Month 12 | 1.56 (37.898) | 25.75 (46.715)
  Septal: Month 6 | 6.40 (33.550) | 9.68 (38.060)
  Septal: Month 12: number analyzed (Participants) | 10 | 13
  Septal: Month 12 | 8.87 (32.843) | 17.17 (39.263)

30. Other Pre Specified Outcome: Change From Baseline in Performance of the Upper Limb (PUL) Overall Score (Excluding Shoulder) at Month 6 and 12
Description: The PUL Scale consists of an entry item to define the starting functional level and 21 items subdivided into shoulder level (4 items), middle level (9 items), and distal level (8 items) dimensions. Each dimension was scored separately with a maximum score of 16 for shoulder level, 34 for middle level, and 24 for distal level. The total score is calculated by the sum of all the scores of the three subscales (excluding the shoulder dimension) and ranged from 0 to 58. Higher scores indicated improvement and lower scores indicated severity. Change from Baseline in PUL overall score (excluding shoulder) at Month 6 and 12 is reported in this outcome measure.
Time Frame: Baseline, Month 6 and 12
Population: Analysis was performed on mITT population. Here, and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
score on a scale
  Month 6: number analyzed (Participants) | 11 | 12
  Month 6 | -1.8 (4.38) | -0.3 (2.90)
  Month 12: number analyzed (Participants) | 9 | 12
  Month 12 | -1.2 (2.64) | 1.3 (6.12)

31. Other Pre Specified Outcome: Change From Baseline in Performance of the Upper Limb (PUL) Overall Score (Including Shoulder) at Month 6 and 12
Description: The PUL Scale consists of an entry item to define the starting functional level and 21 items subdivided into shoulder level (4 items,), middle level (9 items), and distal level (8 items) dimensions. Each dimension was scored separately with a maximum score of 16 for shoulder level, 34 for middle level, and 24 for distal level. The total score is calculated by the sum of all the scores of the three subscales (including the shoulder dimension) and ranged from 0 to 74. Higher scores over time indicate improvement and lower scores indicated severity. Change from Baseline in PUL overall score (including shoulder) at Month 6 and 12 is reported in this outcome measure.
Time Frame: Baseline, Month 6 and 12
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 6 | 3
score on a scale
  Month 6 | 0.3 (2.16) | -3.7 (4.04)
  Month 12 | -1.8 (3.60) | -4.0 (0.00)

32. Other Pre Specified Outcome: Change From Baseline in Peak Expiratory Flow (PEF) at Month 6 and 12
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: liter per second
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
liter per second
  Month 6: number analyzed (Participants) | 10 | 13
  Month 6 | -0.028 (0.7839) | -0.086 (1.2507)
  Month 12: number analyzed (Participants) | 10 | 11
  Month 12 | 0.095 (0.6134) | -0.101 (1.4427)

33. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Peak Expiratory Flow at Month 6 and 12
Description: Percent predicted PEF is a measure of the maximal or peak flow produced during an exhalation with maximal effort and, as such, is the most effort-dependent measure of lung function.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent predicted PEF
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent predicted PEF
  Month 6: number analyzed (Participants) | 10 | 13
  Month 6 | -3.2 (10.45) | -4.8 (17.53)
  Month 12: number analyzed (Participants) | 10 | 11
  Month 12 | -4.5 (8.90) | -7.1 (20.46)

34. Other Pre Specified Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Month 6 and 12
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by a spirometer.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
mL
  Month 6: number analyzed (Participants) | 10 | 13
  Month 6 | 0.020 (0.3516) | -0.007 (0.2493)
  Month 12: number analyzed (Participants) | 10 | 11
  Month 12 | 0.121 (0.3145) | -0.015 (0.2297)

35. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second at Month 6 and 12
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by a spirometer.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent predicted FEV1
  Month 6: number analyzed (Participants) | 10 | 13
  Month 6 | -1.6 (13.88) | -3.2 (7.82)
  Month 12: number analyzed (Participants) | 10 | 11
  Month 12 | -2.1 (14.15) | -4.3 (7.47)

36. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity Level at Month 6 and 12
Description: FVC was the total amount of air exhaled from the lungs during the lung function test measured by spirometer.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
percent predicted FVC
  Month 6: number analyzed (Participants) | 10 | 13
  Month 6 | -3.6 (14.28) | -3.1 (8.06)
  Month 12: number analyzed (Participants) | 10 | 11
  Month 12 | -6.0 (12.13) | -4.4 (7.17)

37. Other Pre Specified Outcome: Change From Baseline in Forced Vital Capacity (FVC) Levels at Month 6 and 12
Description: FVC was the total amount of air exhaled from the lungs during the lung function test measured by spirometer.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
mL
  Month 6: number analyzed (Participants) | 10 | 13
  Month 6 | -0.028 (0.2732) | 0.007 (0.3101)
  Month 12: number analyzed (Participants) | 10 | 11
  Month 12 | 0.000 (0.2240) | -0.014 (0.2383)

38. Other Pre Specified Outcome: Change From Baseline in Forced Expiratory Flow at 25-75% of FVC (FEF25-75%) at Month 6 and 12
Description: Forced Expiratory Flow (FEF) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEF25-75% is defined as the mean forced expiratory flow between the 25% and 75% of the FVC (total amount of air exhaled from the lungs during the lung function test).
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: liter per second
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 12
liter per second
  Month 6: number analyzed (Participants) | 10 | 12
  Month 6 | 0.097 (1.0146) | 0.139 (0.9876)
  Month 12: number analyzed (Participants) | 10 | 10
  Month 12 | 0.437 (0.7612) | 0.166 (1.0708)

39. Other Pre Specified Outcome: Change From Baseline in Percent Predicted Forced Expiratory Flow at 25-75% of FVC at Month 6 and 12
Description: FEF is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEF25-75% is defined as the mean forced expiratory flow between the 25% and 75% of the FVC (total amount of air exhaled from the lungs during the lung function test).
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent predicted FEF
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 12
percent predicted FEF
  Month 6: number analyzed (Participants) | 10 | 12
  Month 6 | 0.2 (23.05) | 1.1 (23.65)
  Month 12: number analyzed (Participants) | 10 | 10
  Month 12 | 5.6 (20.34) | 0.9 (26.24)

40. Other Pre Specified Outcome: Change From Baseline in Forced Expiratory Time (FET) at Month 6 and 12
Description: FET is defined as the time taken for an individual to complete a forceful exhalation after maximal inspiration. FET is measured by asking the subject to take a deep breath and blow it all out as fast as possible.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
seconds
  Month 6: number analyzed (Participants) | 8 | 9
  Month 6 | -0.433 (1.5197) | 0.547 (2.6335)
  Month 12: number analyzed (Participants) | 9 | 7
  Month 12 | 0.086 (0.6403) | 0.181 (2.5598)

41. Other Pre Specified Outcome: Change From Baseline in Six-Minute Walk Test at Month 6 and 12
Description: The six-minute walk test measures the distance a participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the participant to walk as far as possible in six minutes. The participant is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. The total distance walked, in meters, was recorded for each participant. Longer distances indicate better outcomes.
Time Frame: Baseline, Month 6 and 12
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 2 | 2
meters
  Month 6 | -9.0 (2.83) | -68.5 (21.92)
  Month 12 | -8.5 (0.71) | -117.0 (4.24)

42. Other Pre Specified Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Total Summary Score - Participant Responses at Month 6 and 12
Description: The PedsQL-Duchenne muscular dystrophy (DMD) module consists of 18 items and comprised of 4 domains: Daily Activities, Treatment Barriers, Worry, Communication. Items are reverse scored and linearly transformed to a 0-100 scale. The overall range for total PedsQL score (18 items; mean of all items) was 0 (improvement) to 100 (severity). Decreasing scores over time indicate improvement. Change From Baseline in PedsQL total summary score- participant responses at Month 6 and 12 was reported in this outcome measure.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
score on a scale
  Month 6: number analyzed (Participants) | 10 | 13
  Month 6 | -9.83 (10.507) | 3.64 (16.225)
  Month 12: number analyzed (Participants) | 9 | 13
  Month 12 | -11.24 (11.293) | 4.28 (16.455)

43. Other Pre Specified Outcome: Change From Baseline in Pediatric Quality of Life Inventory Total Summary Score - Parent Responses at Month 6 and 12
Description: The PedsQL-Duchenne muscular dystrophy (DMD) module consists of 18 items and comprised of 4 domains: Daily Activities, Treatment Barriers, Worry, Communication. Items are reverse scored and linearly transformed to a 0-100 scale. The overall range for total PedsQL score (18 items; mean of all items) was 0 (improvement) to 100 (severity). Decreasing scores over time indicate improvement. Change From Baseline in PedsQL total summary score- parent responses at Month 6 and 12 was reported in this outcome measure.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
score on a scale
  Month 6: number analyzed (Participants) | 10 | 13
  Month 6 | -1.40 (13.495) | -0.21 (17.334)
  Month 12: number analyzed (Participants) | 10 | 13
  Month 12 | -6.69 (7.627) | -0.43 (19.429)

44. Other Pre Specified Outcome: Change From Baseline in Pediatric Outcomes Data Collection Instrument (PODCI) Score - Parent Responses at Month 6 and 12
Description: The PODCI consists of 83 items and 5 core scales: Upper Extremity and Physical Function, Transfer/Basic Mobility, Sports/Physical Functioning, Pain/Comfort, and Happiness; a Global Functioning Scale. The Global Functioning Scale is the mean of the mean scores from 4 of the 5 core scales (all except the happiness core scale). The Global Functioning Scale and each of the core scales were standardized so that a score of "0" represents a poor outcome/worse health, while "100" is the best possible outcome/best health (i.e., complete range of each score is 0 to 100, with higher scores representing better functioning).
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
score on a scale
  Upper Extremity and Physical Function: Month 6: number analyzed (Participants) | 10 | 13
  Upper Extremity and Physical Function: Month 6 | 3.9 (9.81) | -2.5 (13.17)
  Upper Extremity and Physical Function: Month 12: number analyzed (Participants) | 10 | 13
  Upper Extremity and Physical Function: Month 12 | -3.9 (5.51) | -2.5 (12.36)
  Transfer and Basic Mobility: Month 6: number analyzed (Participants) | 10 | 13
  Transfer and Basic Mobility: Month 6 | -2.8 (9.69) | -1.2 (6.19)
  Transfer and Basic Mobility: Month 12: number analyzed (Participants) | 10 | 12
  Transfer and Basic Mobility: Month 12 | -7.9 (8.91) | -2.3 (8.71)
  Sports/Physical Functioning: Month 6: number analyzed (Participants) | 10 | 13
  Sports/Physical Functioning: Month 6 | 0.0 (7.48) | -1.6 (10.21)
  Sports/Physical Functioning: Month 12: number analyzed (Participants) | 10 | 13
  Sports/Physical Functioning: Month 12 | -0.9 (16.35) | -2.9 (9.60)
  Pain/Comfort: Month 6: number analyzed (Participants) | 10 | 13
  Pain/Comfort: Month 6 | 8.6 (22.38) | 2.0 (11.73)
  Pain/Comfort: Month 12: number analyzed (Participants) | 10 | 13
  Pain/Comfort: Month 12 | 1.8 (22.58) | -1.5 (20.39)
  Happiness: Month 6: number analyzed (Participants) | 10 | 13
  Happiness: Month 6 | -2.5 (16.20) | 4.2 (13.20)
  Happiness: Month 12: number analyzed (Participants) | 10 | 13
  Happiness: Month 12 | -16.5 (14.54) | 8.1 (10.71)
  Global Function: Month 6: number analyzed (Participants) | 10 | 13
  Global Function: Month 6 | 2.6 (9.00) | -0.8 (8.01)
  Global Function: Month 12: number analyzed (Participants) | 10 | 13
  Global Function: Month 12 | -2.5 (8.46) | -2.1 (8.15)

45. Other Pre Specified Outcome: Change From Baseline in Pediatric Outcomes Data Collection Instrument (PODCI) Score - Participant Responses at Month 6 and 12
Description: as for outcome 44
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
score on a scale
  Upper Extremity and Physical Function: Month 6: number analyzed (Participants) | 10 | 13
  Upper Extremity and Physical Function: Month 6 | -3.7 (6.04) | -3.2 (8.84)
  Upper Extremity and Physical Function: Month 12: number analyzed (Participants) | 9 | 13
  Upper Extremity and Physical Function: Month 12 | -5.1 (8.82) | -1.8 (14.25)
  Transfer and Basic Mobility: Month 6: number analyzed (Participants) | 10 | 13
  Transfer and Basic Mobility: Month 6 | -5.9 (8.44) | -4.2 (6.37)
  Transfer and Basic Mobility: Month 12: number analyzed (Participants) | 9 | 13
  Transfer and Basic Mobility: Month 12 | -11.2 (9.86) | -2.7 (9.70)
  Sports/Physical Functioning: Month 6: number analyzed (Participants) | 10 | 13
  Sports/Physical Functioning: Month 6 | -9.9 (10.89) | -2.5 (7.34)
  Sports/Physical Functioning: Month 12: number analyzed (Participants) | 9 | 13
  Sports/Physical Functioning: Month 12 | -11.4 (12.66) | -6.8 (13.06)
  Pain/Comfort: Month 6: number analyzed (Participants) | 10 | 13
  Pain/Comfort: Month 6 | 6.4 (16.75) | 1.0 (13.34)
  Pain/Comfort: Month 12: number analyzed (Participants) | 9 | 13
  Pain/Comfort: Month 12 | 6.2 (24.13) | 2.2 (13.03)
  Happiness: Month 6: number analyzed (Participants) | 10 | 13
  Happiness: Month 6 | 2.0 (14.94) | 2.3 (31.07)
  Happiness: Month 12: number analyzed (Participants) | 9 | 13
  Happiness: Month 12 | -8.3 (21.21) | 12.3 (27.96)
  Global Function: Month 6: number analyzed (Participants) | 10 | 13
  Global Function: Month 6 | -3.3 (4.00) | -2.3 (4.46)
  Global Function: Month 12: number analyzed (Participants) | 9 | 13
  Global Function: Month 12 | -5.4 (4.59) | -2.2 (5.73)

46. Other Pre Specified Outcome: Change From Baseline in Duchenne Muscular Dystrophy Biomarkers at Month 6 and 12
Description: Osteopontin, Cardiac stress biomarker (ST2) and Galectin-3 were DMD biomarkers assessed through serum samples.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Usual Care | CAP-1002
Number analyzed (Participants) | 11 | 13
nanograms per milliliter
  Galectin-3: Month 6: number analyzed (Participants) | 10 | 12
  Galectin-3: Month 6 | 0.368 (1.8119) | -0.175 (2.9025)
  Galectin-3: Month 12: number analyzed (Participants) | 10 | 13
  Galectin-3: Month 12 | 2.958 (4.9781) | 0.829 (1.3238)
  Osteopontin: Month 6: number analyzed (Participants) | 9 | 8
  Osteopontin: Month 6 | 9.238 (24.0751) | 8.051 (14.6530)
  Osteopontin: Month 12: number analyzed (Participants) | 7 | 9
  Osteopontin: Month 12 | 5.400 (31.2415) | 14.868 (18.1615)
  ST2: Month 6: number analyzed (Participants) | 10 | 13
  ST2: Month 6 | 3.99 (15.574) | -9.43 (16.294)
  ST2: Month 12: number analyzed (Participants) | 8 | 10
  ST2: Month 12 | -7.61 (14.928) | -21.10 (19.637)

ADVERSE EVENTS:
Time Frame: Adverse Events data was collected from first infusion up to 12 Month post-infusion
Description: Analysis was performed on safety population.
Arm/Group | Usual Care | CAP-1002
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/12 | 3/13
Other Adverse Events (participants affected / at risk) | 9/12 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=12) | CAP-1002 (N=13)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=12) | CAP-1002 (N=13)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 5 (5)
Atrioventricular Block Second Degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter Site Pain (General disorders) | 0 (0) | 1 (1)
Body Tinea (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (5)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Heart Rate Irregular (Investigations) | 1 (1) | 0 (0)
Monocyte Count Decreased (Investigations) | 1 (1) | 0 (0)
Spirometry abnormal (Investigations) | 0 (0) | 1 (1)
Troponin Increased (Investigations) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 0 (0)
Insulin Resistance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT02485938/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT02485938/SAP_001.pdf